CLINICAL TRIAL: NCT01781962
Title: A Study of Quantitative Assessments of Angle Width in Chinese Patients With Open-angle Glaucoma and/or Ocular Hypertension
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to corporate decision.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 192024-077
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Results first posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Open-Angle Glaucoma (OAG) and/or Ocular Hypertension (OHT) patients.
  Interventions: Other: No Treatment

INTERVENTIONS:
Other: No Treatment — No Treatment was given in this study.

SUMMARY:
This study will assess angle width in Chinese patients with Open-angle Glaucoma and/or Ocular Hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Of Chinese descent
* Open-angle Glaucoma or Ocular Hypertension in each eye

Exclusion Criteria:

* History of a narrow-angle or angle closure glaucoma
* Angle abnormalities in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients with Open-angle Glaucoma and/or Ocular Hypertension
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Beijing, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 206
Completed | 201
Not Completed | 5
Not completed — Other Miscellaneous Reasons | 5

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 206
Age, Customized [Number; unit: Participants]
  <45 years | 111
  45 to 65 years | 71
  >65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 115

OUTCOME MEASURES:

1. Primary Outcome: Anterior Angle Width Using Anterior Segment Optical Coherence Tomography (AS OCT)
Description: The angle width formed between the eye's cornea and iris in both eyes was measured in microns (µm) using AS OCT, a laser-based, noninvasive, diagnostic system providing high-resolution images of the eye.
Time Frame: Day 1
Population: Participants from the Modified Intent-to-treat (mITT) population, all enrolled patients with both gonioscopy and AS OCT measurements, with evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: Eyes
Arm/Group | All Participants
Number analyzed (Participants) | 179
Number analyzed (Eyes) | 330
µm | 638.8 (272.67)

2. Secondary Outcome: Number of Study Eyes in Each Shaffer Grade Using Gonioscopic Lens
Description: The angle width formed between the cornea and iris in both eyes was measured by gonioscopy using Shaffer grading where: grade 4=wide open, grade 3=moderately open, grade 2=moderately narrow, grade 1=very narrow or grade 0=closed. The number of eyes in each Shaffer Grade is reported.
Time Frame: Day 1
Population: Participants from the mITT population, all enrolled patients with both gonioscopy and AS OCT measurements, with data available for this outcome measure.
Measure: Number; unit: eye
Units Other Than Participants: Eyes
Arm/Group | All Participants
Number analyzed (Participants) | 203
Number analyzed (Eyes) | 405
eye
  Grade 1 | 1 (NA)
  Grade 2 | 1 (NA)
  Grade 3 | 34 (334.86)
  Grade 4 | 369 (262.33)

3. Secondary Outcome: Number of Study Eyes in Each Step Grade Using Gonioscopic Lens
Description: The angle width formed between the cornea and iris in both eyes was measured by gonioscopy using Large Step Grading ranging from 1.0 (smallest angle width) to 7.5 (largest angle width) with 0.5 unit intervals where each Large Step unit represented a fixed length of approximately 200 µm. The number of eyes in each Large Step Grade is reported.
Time Frame: Day 1
Population: as for outcome 2
Measure: Number; unit: eye
Units Other Than Participants: Eyes
Arm/Group | All Participants
Number analyzed (Participants) | 203
Number analyzed (Eyes) | 405
eye
  Step Grade 1.0 | 0 (126.92)
  Step Grade 1.5 | 4 (203.66)
  Step Grade 2.0 | 36 (206.72)
  Step Grade 2.5 | 32 (212.36)
  Step Grade 3.0 | 78 (191.87)
  Step Grade 3.5 | 24 (234.94)
  Step Grade 4.0 | 69 (290.20)
  Step Grade 4.5 | 23 (208.44)
  Step Grade 5.0 | 34 (119.57)
  Step Grade 5.5 | 9 (221.46)
  Step Grade 6.0 | 33 (184.16)
  Step Grade 6.5 | 28 (294.97)
  Step Grade 7.0 | 28 (158.44)
  Step Grade 7.5 | 7

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Screening through Day 1 (Up to 5 Weeks)
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/206
Other Adverse Events (participants affected / at risk) | 0/206

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.